CLINICAL TRIAL: NCT04358276
Title: Technology-Enabled Activation of Skin Cancer Screening for Hematopoietic Cell Transplantation Survivors and Their Primary Care Providers (TEACH)
Brief Title: Technology-Enabled Activation of Skin Cancer Screening for Stem Cell Transplant Survivors and Their Primary Care Providers, TEACH Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20096; NCI-2020-01830 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20096 (Other: City of Hope Medical Center); 38249 (Other: National Cancer Institute)
Record Dates: First submitted 2020-04-07; First posted 2020-04-24 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Skin Carcinoma
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods; Physicians; Communication Devices for People with Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group I (PAE) (Experimental): Participants receive a study packet on skin cancer. Participants also receive text messages once every 3 weeks for 9 months.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration; Other: Text Message
- Group II (PAE, physician) (Experimental): Participants receive a study packet on skin cancer. Participants also receive text messages once every 3 weeks for 9 months. Participants' physician receives a letter that describes the educational intervention and encourages them to do a skin examination at next patient visit.
  Interventions: Other: Educational Intervention; Other: Educational Intervention (Physician); Other: Questionnaire Administration; Other: Text Message
- Group III (PAE, physician, dermatoscope) (Experimental): Participants receive a study packet on skin cancer. Participants also receive text messages once every 3 weeks for 9 months. Participants' physician receives a letter that describes the educational intervention and encourages them to do a skin examination at next patient visit. Physicians also receive a free dermatoscope with instructions for uploading images of suspect lesions and attend a 30-minute online course comprising additional descriptions of dermoscopic images for skin cancers and "mimickers" common in hematopoietic stem cell transplantation patients, along with clear instructions for using a dermatoscope and steps to integrate dermoscopy into their practice.
  Interventions: Other: Computer-Assisted Intervention; Device: Dermatoscope; Other: Educational Intervention; Other: Educational Intervention (Physician); Other: Questionnaire Administration; Other: Text Message

INTERVENTIONS:
Other: Computer-Assisted Intervention — Complete online course
  Arms: Group III (PAE, physician, dermatoscope)
Device: Dermatoscope — Receive dermatoscope
  Arms: Group III (PAE, physician, dermatoscope)
Other: Educational Intervention — Receive study packet
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Educational Intervention (Physician) — Receive physician directed letter and educational package
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (PAE, physician); Group III (PAE, physician, dermatoscope)
Other: Questionnaire Administration — Ancillary studies
Other: Text Message — Receive text messages
  Other Names: SMS Text; SMS Text Message; Text

SUMMARY:
This trial studies the impact of a 12-month invention focused on early detection of skin cancer and timely follow up in patients who underwent stem cell transplant and their primary care providers. Some stem cell transplant survivors may develop complications related to the treatment they received. Many of these complications may not be known for years after the treatment and preventive measures can be taken to reduce the chances that a complication will occur and encourage early detection. This study focuses on one complication that stem cell transplant survivors are at high risk of developing - skin cancer. An early diagnosis of skin cancer is important since the cancer is usually smaller, requires less extensive treatments, and has better outcomes. Teaching skin self-examination and encouraging patients to alert doctors to skin changes may provide an important opportunity for early detection of skin cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the impact of patient activation and education (PAE, N=360) alone or with physician activation (PAE+Phys, N=360) on skin cancer screening and health promotion practices at 12 months, measured by percentage of survivors who conduct skin self-exam and receive physician skin exam, and time to detection and diagnosis of suspicious lesions.

II. Among primary care physicians of transplant patients, determine the impact of an e-learning teledermoscopy program compared with provision of print materials for identifying suspect lesions.

OUTLINE: Participants are randomized to 1 of 3 groups.

GROUP I: Participants receive a study packet on skin cancer. Participants also receive text messages once every 3 weeks for 9 months.

GROUP II: Participants receive a study packet on skin cancer. Participants also receive text messages once every 3 weeks for 9 months. Participants' physician receives a letter that describes the educational intervention and encourages them to do a skin examination at next patient visit.

GROUP III: Participants receive a study packet on skin cancer. Participants also receive text messages once every 3 weeks for 9 months. Participants' physician receives a letter that describes the educational intervention and encourages them to do a skin examination at next patient visit. Physicians also receive a free dermatoscope with instructions for uploading images of suspect lesions and attend a 30-minute online course comprising additional descriptions of dermoscopic images for skin cancers and "mimickers" common in hematopoietic stem cell transplantation patients, along with clear instructions for using a dermatoscope and steps to integrate dermoscopy into their practice.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone autologous or allogeneic hematopoietic stem cell transplantation (HCT) at City of Hope (COH)
* Are 2 years (yrs) to 5 yrs (+/- 3 months [m]) after HCT
* Have seen a primary care provider (PCP) in the previous 12 m (expected > 95% of all eligible) or planning to do so in next 12 m
* Have a mobile phone with the ability to receive text messages
* Can fluently read and write in English or Spanish
* Can understand and sign the study-specific Informed Consent Form (ICF)

Exclusion Criteria:

* Patients who have evidence of active hematologic malignancy or acute illness that would limit study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Impact of patient activation and education alone or with physician activation on change in skin cancer screening and health promotion practices | Baseline and 12 months
  Will administer questionnaires at baseline and 12 months to ask about skin examinations performed within the past 12 months. Will use logistic regression to adjust for imbalance in patient characteristics and risk factors. Will also test for group by covariate interactions, depending on group main effect.
Time interval between a participant's first notice of a suspect mole or lesion and the date on which a definitive diagnosis was made | Up to 12 months
  Will be a continuous variable, and will employ a generalized linear model to compare the interval between the two study arms, adjusted for covariates of interest. Will begin with bivariate models to determine potential variables to include in a multivariable regression model. If the group main effect is significant, interactions of the group main effect with other variables will be examined.
Impact of an e-learning teledermoscopy program compared with provision of print materials for identifying suspect lesions | Up to 12 months
  Will compare the group difference in changes in attitude over time, using generalized estimating equation (GEE) for normally distributed data, with a compound symmetry covariance matrix analysis to account for within-physician correlation. Will dichotomize the Likert scale (1-5) response and compare the proportion of primary care physicians (PCPs) reporting a higher (>= 4 versus < 4) level of confidence at 12 months (m) compared to baseline between groups, using the longitudinal binomial GEE model with a compound symmetry covariance structure. Covariate adjustment will be made in these models as necessary.
Economic impact on patients - cost-effectiveness analysis | Up to 12 months
  Evaluated using standard incremental cost-effectiveness analysis methods will be used to assess the impact of assumptions and uncertainty on results and conclusions.
Economic impact on patients - sensitivity analysis | Up to 12 months
  Evaluated using standard incremental sensitivity analysis will be used to assess the impact of assumptions and uncertainty on results and conclusions.
Downstream costs | Up to 12 months
  Will estimate the cost per additional self skin exam completed and the cost per additional PCP exam completed, comparing the two intervention arms.

CONTACTS AND LOCATIONS:
Overall Officials: Saro H Armenian, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Armenian SH, Lindenfeld L, Iukuridze A, Echevarria M, Bebel S, Coleman C, Nakamura R, Abdullah F, Modi B, Oeffinger KC, Emmons KM, Marghoob AA, Geller AC. Technology-enabled activation of skin cancer screening for hematopoietic cell transplantation survivors and their primary care providers (TEACH). BMC Cancer. 2020 Aug 3;20(1):721. doi: 10.1186/s12885-020-07232-2. PMID 32746799

DOCUMENTS (1):
  • Informed Consent Form (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04358276/ICF_000.pdf